CLINICAL TRIAL: NCT02868918
Title: Clinical and Radiographical Evaluation of New Bioactive Dentine Substitute (Biodentine) Versus Glass Ionomer Cement in Treatment of Very Deep Carious Lesions -Randomized Clinical Trial
Brief Title: Evaluation of Biodentine Versus Glass Ionomer Cement in Treatment of Very Deep Carious Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Magdy Moustafa, Assistant lecturer , Conservative Dentistry Department, Faculty of Oral & Dental Medicine Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CEBD-CU-2016-08-174
Record Dates: First submitted 2016-08-06; First posted 2016-08-16 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Deep Caries
MeSH Terms: interventions — tricalcium silicate; Glass Ionomer Cements; fuji IX; Radiographic Image Enhancement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- biodentine (Experimental): bioactive dentin substitute used to act like natural dentin in insulating the pulp against external stimuli intervention
  Interventions: Drug: biodentine; Device: DigoraH optium
- glass ionomer cement (Active Comparator): high viscosity glass ionomer used as a base material comparator other name : - fuji ix
  Interventions: Drug: glass ionomer cement; Device: DigoraH optium

INTERVENTIONS:
Drug: biodentine — tricalcium silicate cement used to replace the carious dentin
  Other Names: tricalcium silicate
  Arms: biodentine
Drug: glass ionomer cement — high viscosity glass ionomer used as a base material
  Other Names: Fuji ix
  Arms: glass ionomer cement
Device: DigoraH optium — digital Xray for follow up
  Other Names: digital radiography

SUMMARY:
The aim of this study is to compare the effect of new bioactive dentine substitute (Biodentine) versus glass ionomer cement in very deep carious lesions clinically and radiographically using digital radiography in the terms of postoperative pain and biocompatibility to the pulp.

DETAILED DESCRIPTION:
Roles and responsibilities:

* Omnia Magdy Moustafa (O.M.) Operator, data entry & corresponding author; Assistant lecturer ,
* Mohmed Riad Farid (M.R.) Main supervisor, data monitoring & auditing; Professor, Conservative Dentistry
* Rasha Raffat (R.R.) Co-supervisor, data entry & auditing; Lecturer, Conservative Dentistry Department
* Amir Hafez Ibrahim (A.H.), *Mohamed Refaat El-Bialy (M.E.) (A.H) Lecturer, Conservative Dentistry Department, Faculty of Oral & Dental Medicine Cairo University,(M.E.) Assistant lecturer , Conservative Dentistry Department, Faculty of Oral & Dental Medicine Cairo University outcome assessors and data collection.
* Omar Shalaan (O.S.) Demonstrator, Conservative Dentistry Department, Faculty of Oral & Dental Medicine Cairo University, for baseline data collection, recruitment, sequence generation, allocation concealment, patient retention and taking participants consents.

Interventions:

* Pre-operative clinical assessment :

  1. Thermal testing using Refrigerant spray
  2. percussion test
  3. Palpation and clinical examination
  4. peri-apical radiographs using digital radiograph
* Caries removal procedure:

Local anesthesia will be given to the patient then complete isolation to the tooth using rubber dame the operator O.M. will open the enamel Then in caries removal from the walls carbon-steel rose-head bur. Finally the deeper caries will be removed using spoon excavator

* Intervention : Biodentine™ (Septodont, St. Maur-des-Fossés, France) The material will be applied according to manufacturer instructions
* Comparator: GC Fuji IX GP (GC America Inc, Alsip, IL, USA) The material will be applied according to manufacturer instructions
* Final restoration application:

Filtek™ Z250 Universal Restorative (3M Canada, London, Ontario Canada)

-Adhesive system: Scotchbond Universal Etchant (3M ESPE, St. Paul MN, USA) & Single Bond Universal adhesive (3M ESPE, St. Paul MN, USA).

* The material will be applied according to manufacturer instruction

ELIGIBILITY:
Inclusion Criteria:

1. Patients male or female older than 18 y in good general health
2. A minimum of 1 deep carious lesion penetrating three-quarters or more into the dentine as identified with the periapical (PA) radiograph; Clinically according to International Caries Detection and Assessment System (ICDAS II) score 4
3. Clinical symptoms of reversible pulpitis
4. Positive pulp response to electric pulp test or thermal stimulation
5. No PA changes viewed on PA radiograph

Exclusion Criteria:

1. Clinical symptoms of irreversible pulpitis requiring endodontic treatment
2. Presence of fistulas or swelling
3. Mobile teeth or tenderness to percussion
4. Anterior teeth with aesthetic concerns
5. Pregnant women, in view of requirements for radiographs
6. Patients younger than 18 y
7. Patients unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
postoperative hypersensitivity using yes or no questionnaire | 6 months

SECONDARY OUTCOMES:
Biocompatibility of biodentine using digital X-ray | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkhadem, PhD, Study Chair — Cairo University
Locations (1):
- Omnia Magdy, Cairo, Egypt